CLINICAL TRIAL: NCT01463683
Title: A Study in Healthy Japanese Young Adults to Assess the Safety, Tolerability, and Immunogenicity of HEPTAVAX-II Manufactured Using a Modified Process
Brief Title: Modified Process Hepatitis B Vaccine in Japanese Young Adults (V232-062)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V232-062
Record Dates: First submitted 2011-10-28; First posted 2011-11-02 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Recombivax HB; Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- V232-2XP SC (Experimental): 2XP HEPTAVAX™-II vaccine 10 mcg in 0.5 mL subcutaneous injection on Day 1, Month 1, and Month 6
  Interventions: Biological: 2XP HEPTAVAX™-II SC
- V232-1XP SC (Active Comparator): 1XP HEPTAVAX™-II vaccine 10 mcg in 0.5 mL subcutaneous injection on Day 1, Month 1, and Month 6
  Interventions: Biological: 1XP HEPTAVAX™-II SC
- V232-2XP IM (Experimental): 2XP HEPTAVAX™-II vaccine 10 mcg in 0.5 mL intramuscular injection on Day 1, Month 1, and Month 6
  Interventions: Biological: 2XP HEPTAVAX™-II IM

INTERVENTIONS:
Biological: 2XP HEPTAVAX™-II SC
  Other Names: RECOMBIVAX HB; HBVAXPRO
  Arms: V232-2XP SC
Biological: 1XP HEPTAVAX™-II SC
  Other Names: RECOMBIVAX HB; HBVAXPRO
  Arms: V232-1XP SC
Biological: 2XP HEPTAVAX™-II IM
  Arms: V232-2XP IM

SUMMARY:
This is a study to evaluate immunogenicity, safety, and tolerability of 2XP HEPTAVAX™-II compared with the 1XP HEPTAVAX™-II in healthy Japanese young adults.

DETAILED DESCRIPTION:
2XP HEPTAVAX™-II is manufactured using a modified process in which the composition of the amorphous aluminum hydroxyphosphate sulfate adjuvant has been modified by increasing the phosphate content by approximately 2-fold. Thus the modified process HEPTAVAX™-II is referred to as 2XP HEPTAVAX™-II.

ELIGIBILITY:
Inclusion Criteria:

To receive the first study vaccination, Participants should meet all inclusion criteria.

* Participants provide written informed consent for the trial. The Participant may also provide consent for Future Biomedical Research. However, the Participant may participate in the main trial without participating in Future Biomedical Research.
* Participant is Japanese male or female, between 20 to 35 years of age on the day of the first study vaccination.
* Participant is determined to be in general good health based on the medical history taken on Day 1 prior to receiving the first injection of the vaccine. Any underlying chronic illness must be documented to be in stable condition.
* For females, a negative urine pregnancy test just prior to vaccination on Day 1.

Exclusion Criteria:

To receive the first study vaccination, Participants should not have any exclusion criteria. For items with an asterisk (*), if the Participant meets these exclusion criteria, the visit may be rescheduled for a time when these criteria are not met.

* Participant has a history of previous hepatitis B infection.
* Participant has a history of vaccination with any hepatitis B vaccine.
* *Participant has a recent (≤72 hours) history of febrile illness (oral temperature ≥ 37.8°C).
* Participant has a known or suspected hypersensitivity to any component of HEPTAVAX™-II vaccine and latex (e.g., aluminum, yeast).
* Participant has a recent administration (within 3 months prior to first injection with the study vaccine) of hepatitis B immune globulin (HBIG), serum immune globulin, or any other blood-derived product, or is expected to require such blood-derived products during the study.
* *Participant has received licensed inactivated vaccines within 14 days prior or licensed live vaccines within 28 days prior to first injection with the study vaccine.
* Participant has received investigational drugs or other investigational vaccines within 3 months prior to first injection with the study vaccine.
* Use of immunosuppressive therapy. Participants on corticosteroids should be excluded if they are receiving or are expected to receive, in the period from 4 weeks prior to enrollment until 6 weeks post vaccination, systemic doses greater than required for physiological replacement, i.e., >5 mg of prednisone (or equivalent) per day for >2 weeks (except for use of topical or inhalation steroid therapy).
* Pregnant women, nursing mothers, and women planning to become pregnant within the study period. Women of childbearing age should employ an acceptable method of contraception during the study (e.g., condom, diaphragm, oral contraceptive, Intrauterine Device (IUD), or hormonal implants are considered acceptable).
* Participant has any condition, which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* Participant has a coagulation disorder contraindicating intramuscular injection.
* Participant has immunocompromised condition (such as Human Immunodeficiency Virus (HIV) positive, leukemia, lymphoma, other cancers or disorders).

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 722 (Actual)
Dates: Start 2011-11-29 (Actual); Primary Completion 2012-11-06 (Actual); Study Completion 2012-11-06 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kishino H, Takahashi K, Sawata M, Tanaka Y. Immunogenicity, safety, and tolerability of a recombinant hepatitis B vaccine manufactured by a modified process in healthy young Japanese adults. Hum Vaccin Immunother. 2018 Jul 3;14(7):1773-1778. doi: 10.1080/21645515.2018.1452578. Epub 2018 Apr 12. PMID 29553862

RESULTS

PARTICIPANT FLOW:
Groups:
- V232-2XP Subcutaneous (SC): 2XP HEPTAVAX™-II vaccine 0.5 mL subcutaneous injection on Day 1, Month 1, and Month 6
- V232-1XP SC: 1XP HEPTAVAX™-II vaccine 0.5 mL subcutaneous injection on Day 1, Month 1, and Month 6
- V232-2XP Intramuscular (IM): 2XP HEPTAVAX™-II vaccine 0.5 mL intramuscular injection on Day 1, Month 1, and Month 6
Period: Overall Study
Arm/Group | V232-2XP Subcutaneous (SC) | V232-1XP SC | V232-2XP Intramuscular (IM)
Started | 309 | 309 | 104
Received Vaccination 1 (Day 1) | 309 | 308 | 104
Received Vaccination 2 (Month 1) | 302 | 300 | 103
Received Vaccination 3 (Month 6) | 290 | 281 | 93
Completed | 290 | 278 | 93
Not Completed | 19 | 31 | 11
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lost to Follow-up | 10 | 9 | 7
Not completed — Physician Decision | 0 | 3 | 1
Not completed — Pregnancy | 2 | 2 | 1
Not completed — Withdrawal by Subject | 5 | 17 | 2

BASELINE CHARACTERISTICS:
Groups:
- V232-2XP SC: 2XP HEPTAVAX™-II vaccine 0.5 mL subcutaneous injection on Day 1, Month 1, and Month 6
- V232-2XP IM: 2XP HEPTAVAX™-II vaccine 0.5 mL intramuscular injection on Day 1, Month 1, and Month 6
- Total: Total of all reporting groups
Arm/Group | V232-2XP SC | V232-1XP SC | V232-2XP IM | Total
Number analyzed (Participants) | 309 | 308 | 104 | 721
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.3 (4.7) | 26.8 (4.6) | 26.9 (4.9) | 27.1 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 144 | 48 | 361
  Male | 140 | 164 | 56 | 360

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Receiving Subcutaneous Vaccination Who Achieved Seroprotection
Description: Blood samples were collected for anti-hepatitis B antibody assays. Seroprotection was defined as ≥10 mIU/mL anti-hepatitis B antibody.
Time Frame: Month 7
Population: The per protocol population consisted of all randomized participants who met enrollment criteria, did not violate the protocol, were seronegative at Baseline, and had vaccination and blood collection. Seroprotection was evaluated only for participants receiving vaccine subcutaneously; intramuscular vaccination was evaluated for safety only.
Measure: Number; unit: Percentage of participants
Arm/Group | V232-2XP SC | V232-1XP SC
Number analyzed (Participants) | 247 | 217
Percentage of participants | 90.1 | 82.5
Statistical Analysis 1: Comparison: V232-2XP SC vs V232-1XP SC; Test type: Non-Inferiority or Equivalence — Incidence of seroprotection with V232-2XP SC is non-inferior to V232-1XP SC if the lower bound of the 95% confidence interval of the difference is greater than -10%; Miettinen & Nurminen; Difference in percentage of participants = 7.6, 95% CI 2-sided [1.9 to 13.6]

2. Primary Outcome: Percentage of Participants With Injection-site Adverse Events
Description: Participants were evaluated for injection-site adverse events using MedDRA version 15.1
Time Frame: Up to 15 days after each vaccination
Population: All randomized participants who received at least 1 vaccination were included in the analysis
Measure: Number; unit: Percentage of participants
Arm/Group | V232-2XP SC | V232-1XP SC | V232-2XP IM
Number analyzed (Participants) | 309 | 308 | 104
Percentage of participants | 76.4 | 71.4 | 65.4
Statistical Analysis 1: Comparison: V232-2XP SC vs V232-1XP SC; Test type: Superiority or Other; p = 0.162, Miettinen & Nurminen; Difference in percentage of participants = 4.9, 95% CI 2-sided [-2.0 to 11.9]
Statistical Analysis 2: Comparison: V232-2XP SC vs V232-2XP IM; Test type: Superiority or Other; p = 0.028, Miettinen & Nurminen; Difference in percentage of participants = 11.0, 95% CI 2-sided [1.1 to 21.6]
Statistical Analysis 3: Comparison: V232-1XP SC vs V232-2XP IM; Test type: Superiority or Other; p = 0.246, Miettinen & Nurminen; Difference in percentage of participants = 6.0, 95% CI 2-sided [-4.0 to 16.8]

3. Primary Outcome: Percentage of Participants With Pyrexia Adverse Events
Description: Participants were evaluated for pyrexia adverse events using MedDRA version 15.1. Pyrexia (fever) was defined as an oral temperature ≥37.8°C ( ≥100.0°F).
Time Frame: Up to 15 days after each vaccination
Population: All randomized participants who received at least 1 vaccination were included in the analysis
Measure: Number; unit: Percentage of participants
Arm/Group | V232-2XP SC | V232-1XP SC | V232-2XP IM
Number analyzed (Participants) | 309 | 308 | 104
Percentage of participants | 3.2 | 3.9 | 4.8
Statistical Analysis 1: Comparison: V232-2XP SC vs V232-1XP SC; Test type: Superiority or Other; p = 0.659, Miettinen & Nurminen; Difference in percentage of participants = -0.7, 95% CI 2-sided [-3.8 to 2.4]
Statistical Analysis 2: Comparison: V232-2XP SC vs V232-2XP IM; Test type: Superiority or Other; p = 0.459, Miettinen & Nurminen; Difference in percentage of participants = -1.6, 95% CI 2-sided [-7.7 to 2.2]
Statistical Analysis 3: Comparison: V232-1XP SC vs V232-2XP IM; Test type: Superiority or Other; p = 0.686, Miettinen & Nurminen; Difference in percentage of participants = -0.9, 95% CI 2-sided [-7.1 to 3.0]

ADVERSE EVENTS:
Time Frame: Serious adverse events: up to Month 7; non-serious adverse events: up to 14 days after each vaccination
Description: The analysis population for adverse events was participants who received at least 1 vaccination
Arm/Group | V232-2XP SC | V232-1XP SC | V232-2XP IM
Serious Adverse Events (participants affected / at risk) | 1/309 | 2/308 | 0/104
Other Adverse Events (participants affected / at risk) | 239/309 | 225/308 | 69/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V232-2XP SC (N=309) | V232-1XP SC (N=308) | V232-2XP IM (N=104)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V232-2XP SC (N=309) | V232-1XP SC (N=308) | V232-2XP IM (N=104)
Injection-site erythema (General disorders) | 172 (294) | 152 (288) | 26 (40)
Injection-site pain (General disorders) | 216 (441) | 194 (400) | 62 (120)
Injection-site pruritus (General disorders) | 50 (75) | 54 (81) | 5 (6)
Injection-site swelling (General disorders) | 165 (278) | 149 (253) | 26 (39)
Nasopharyngitis (Infections and infestations) | 12 (12) | 12 (12) | 7 (7)
Headache (Nervous system disorders) | 21 (29) | 20 (28) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.